CLINICAL TRIAL: NCT02318992
Title: Fresh, Frozen or Lyophilized Fecal Microbiota Transplantation for Multiple Recurrent C. Difficile Associated Diarrhea
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Zhi-Dong Jiang, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC-SPH-13-0119
Expanded Access: NCT03786900 (Available)
Record Dates: First submitted 2014-12-09; First posted 2014-12-18 (Estimated); Results first posted 2019-05-13 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Recurrent C. Difficile Associated Diarrhea
MeSH Terms: interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Fecal Microbiota_Fresh (Active Comparator): Donor stool (greater than 150 grams) was collected <4 hours prior to the procedure and then mixed in a homogenizer with 1500 milliliters (mL) (1:10 dilution) sterilized 0.9% sodium chloride (NaCl) in a large sterilized suction canister until a smooth consistency was reached. The suspension was filtered using a coffee filter twice. The microbiota suspension (250mL) was used within 2 hours of preparation (Fresh).
  Interventions: Biological: Fecal Microbiota
- Fecal Microbiota_Frozen (Active Comparator): Donor stool (greater than 150 grams) was collected <4 hours prior to the procedure and then mixed in a homogenizer with 1500 milliliters (mL) (1:10 dilution) sterilized 0.9% NaCl in a large sterilized suction canister until a smooth consistency was reached. The suspension was filtered using a coffee filter twice. The microbiota suspension (250mL) was kept at -80 degrees Celsius (C) freezer labeled with identity (ID) and expiration date which was 6 months after preparation day (Frozen).
  Interventions: Biological: Fecal Microbiota
- Fecal Microbiota_Lyophilized (Active Comparator): Donor stool (greater than 150 grams) was collected <4 hours prior to the procedure and then mixed in a homogenizer with 1500 milliliters (mL) (1:10 dilution) sterilized 0.9% NaCl in a large sterilized suction canister until a smooth consistency was reached. The suspension was filtered using a coffee filter twice. The microbiota suspension (250mL) was starting lyophilization process within 30 minutes after completion of stool filtration (Lyophilized). Lyophilized microbiota products were kept at 4 degrees celsius (C) and were used within 6 months after preparation day.
  Interventions: Biological: Fecal Microbiota

INTERVENTIONS:
Biological: Fecal Microbiota — Fecal Microbiota will be delivered via colonoscopy.

SUMMARY:
The objective of the study is to investigate the efficacy of fresh, frozen or lyophilized fecal microbiota transplantation (FMT) via colonoscopy in patients with recurrent C. difficile associated diarrhea (RCDAD). Frozen, lyophilized or fresh fecal microbiota transplantation (FMT) inoculum will be generated from well-screened healthy volunteer donors of ≥150 gram/sample. Delivery of FMT will be performed colonoscopically. Fecal samples from donors and recipients will be saved for later metagenomic studies to characterize the microbiome of the gut in patients before and after FMT.

ELIGIBILITY:
Inclusion Criteria:

Recipients

* Male and female patients ≥ 18 years of age
* Sexually active male and female patients of child-bearing potential must agree to use an effective method of birth control during the treatment and follow-up period
* Female patients of child-bearing potential must have a negative pregnancy test in the 72 hours before the procedure
* Required to sign an informed consent form
* Deemed likely to survive for ≥ 3 months after enrolment
* Diagnosis of ≥ 3 recurrent CDAD (RCDAD) bouts in outpatients or ≥ 2 bouts of CDAD in an inpatient without other explanation for diarrhea and with ≥ 2 positive fecal tests for C. difficile toxin
* Referred by subjects attending physician who will provide non-transplant care for the subject and follow up at 1, 7, 14, 30 days after FMT
* Received at least one course of adequate antibiotic therapy for CDAD (≥ 10 days of vancomycin at a dose of ≥125 mg four times per day, ≥ 10 days of metronidazole at a dose of 500mg three times per day or fidaxomixin 200mg twice a day for 10 days
* Anti-Clostridium difficile infection (CDI) antibiotic treatment stopped 2-4 days before the transplantation

Donors

* Able to provide and sign informed consent
* Able to complete and sign the donor questionnaire
* Able to adhere to fecal transplantation stool collection requirements

Exclusion Criteria:

Recipients

* Patients with neutropenia with absolute neutrophil count <0.5 x 109/L
* Evidence of toxic megacolon or gastrointestinal perforation on abdominal x-ray
* Peripheral white blood cell count > 15.0 x 109/L AND temperature > 38.0 °C
* Active gastroenteritis due to Salmonella, Shigella, E. coli 0157:H7, Yersinia or Campylobacter, and Norovirus
* Presence of colostomy
* Unable to tolerate human biotherapy (HBT) for any reason
* Requiring systemic antibiotic therapy for more than 7 days
* Actively taking Saccharomyces boulardii or other probiotic
* Severe underlying disease such that the patient is not expected to survive for one or more years or unstable medical condition requiring daily change in treatments
* Prolonged compromised immunity due to cytotoxic chemotherapy or HIV infection

Donors

* Test positive for any of variables
* History of any type of active cancer or autoimmune disease
* History of risk factors for acquisition of HIV, syphilis, Hepatitis B, Hepatitis C, prion or any neurological disease as determined by the donor questionnaire
* History of gastrointestinal disorder, e.g., inflammatory bowel disease, irritable bowel syndrome, chronic constipation or diarrhea
* Antibiotic use or any systemic immunosuppressive agents in the 3 months prior to stool donation
* Receipt of any type of live vaccine within 3 months prior to stool donation
* Current or previous medical or psychosocial condition
* Body mass index over 30

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Herbert L DuPont, MD, Principal Investigator — The University of Texas Health Science Center, Houston; Zhi-Dong Jiang, MD, Dr.PH, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- University of Texas Health Science Center at Housotn, Houston, Texas, United States

REFERENCES:
- [Background] Jiang ZD, Hoang LN, Lasco TM, Garey KW, Dupont HL. Physician attitudes toward the use of fecal transplantation for recurrent Clostridium difficile infection in a metropolitan area. Clin Infect Dis. 2013 Apr;56(7):1059-60. doi: 10.1093/cid/cis1025. Epub 2012 Dec 7. No abstract available. PMID 23223589
- [Background] Mattila E, Uusitalo-Seppala R, Wuorela M, Lehtola L, Nurmi H, Ristikankare M, Moilanen V, Salminen K, Seppala M, Mattila PS, Anttila VJ, Arkkila P. Fecal transplantation, through colonoscopy, is effective therapy for recurrent Clostridium difficile infection. Gastroenterology. 2012 Mar;142(3):490-6. doi: 10.1053/j.gastro.2011.11.037. Epub 2011 Dec 7. PMID 22155369
- [Background] Hamilton MJ, Weingarden AR, Sadowsky MJ, Khoruts A. Standardized frozen preparation for transplantation of fecal microbiota for recurrent Clostridium difficile infection. Am J Gastroenterol. 2012 May;107(5):761-7. doi: 10.1038/ajg.2011.482. Epub 2012 Jan 31. PMID 22290405
- [Background] Brandt LJ. Fecal transplantation for the treatment of Clostridium difficile infection. Gastroenterol Hepatol (N Y). 2012 Mar;8(3):191-4. No abstract available. PMID 22675283
- [Background] Bakken JS, Borody T, Brandt LJ, Brill JV, Demarco DC, Franzos MA, Kelly C, Khoruts A, Louie T, Martinelli LP, Moore TA, Russell G, Surawicz C; Fecal Microbiota Transplantation Workgroup. Treating Clostridium difficile infection with fecal microbiota transplantation. Clin Gastroenterol Hepatol. 2011 Dec;9(12):1044-9. doi: 10.1016/j.cgh.2011.08.014. Epub 2011 Aug 24. PMID 21871249
- [Background] EISEMAN B, SILEN W, BASCOM GS, KAUVAR AJ. Fecal enema as an adjunct in the treatment of pseudomembranous enterocolitis. Surgery. 1958 Nov;44(5):854-9. No abstract available. PMID 13592638
- [Background] Brandt LJ, Reddy SS. Fecal microbiota transplantation for recurrent clostridium difficile infection. J Clin Gastroenterol. 2011 Nov;45 Suppl:S159-67. doi: 10.1097/MCG.0b013e318222e603. PMID 21992957
- [Background] Borody TJ, Warren EF, Leis S, Surace R, Ashman O. Treatment of ulcerative colitis using fecal bacteriotherapy. J Clin Gastroenterol. 2003 Jul;37(1):42-7. doi: 10.1097/00004836-200307000-00012. PMID 12811208
- [Background] Bennet JD, Brinkman M. Treatment of ulcerative colitis by implantation of normal colonic flora. Lancet. 1989 Jan 21;1(8630):164. doi: 10.1016/s0140-6736(89)91183-5. No abstract available. PMID 2563083
- [Background] Caporaso JG, Lauber CL, Walters WA, Berg-Lyons D, Huntley J, Fierer N, Owens SM, Betley J, Fraser L, Bauer M, Gormley N, Gilbert JA, Smith G, Knight R. Ultra-high-throughput microbial community analysis on the Illumina HiSeq and MiSeq platforms. ISME J. 2012 Aug;6(8):1621-4. doi: 10.1038/ismej.2012.8. Epub 2012 Mar 8. PMID 22402401
- [Background] Edgar RC. Search and clustering orders of magnitude faster than BLAST. Bioinformatics. 2010 Oct 1;26(19):2460-1. doi: 10.1093/bioinformatics/btq461. Epub 2010 Aug 12. PMID 20709691
- [Background] Caporaso JG, Kuczynski J, Stombaugh J, Bittinger K, Bushman FD, Costello EK, Fierer N, Pena AG, Goodrich JK, Gordon JI, Huttley GA, Kelley ST, Knights D, Koenig JE, Ley RE, Lozupone CA, McDonald D, Muegge BD, Pirrung M, Reeder J, Sevinsky JR, Turnbaugh PJ, Walters WA, Widmann J, Yatsunenko T, Zaneveld J, Knight R. QIIME allows analysis of high-throughput community sequencing data. Nat Methods. 2010 May;7(5):335-6. doi: 10.1038/nmeth.f.303. Epub 2010 Apr 11. No abstract available. PMID 20383131

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 79 were enrolled; however only 78 started--this is because one person who enrolled withdrew before treatment initiation due to insurance problem.
Groups:
- Fecal Microbiota_Fresh: Donor stool (greater than 150 grams) was collected <4 hours prior to the procedure and then mixed in a homogenizer with 1500 milliliters (mL) (1:10 dilution) sterilized 0.9% sodium chloride (NaCl) in a large sterilized suction canister until a smooth consistency was reached. The suspension was filtered using a coffee filter twice. The microbiota suspension (250 milliliters (mL)) was used within 2 hours of preparation (Fresh).
  Fecal Microbiota: Fecal Microbiota will be delivered via colonoscopy.
- Fecal Microbiota_Frozen: Donor stool (greater than 150 grams) was collected <4 hours prior to the procedure and then mixed in a homogenizer with 1500 milliliters (mL) (1:10 dilution) sterilized 0.9% sodium chloride (NaCl) in a large sterilized suction canister until a smooth consistency was reached. The suspension was filtered using a coffee filter twice. The microbiota suspension (250mL) was kept at -80 degrees celsius (C) freezer labeled with identity (ID) and expiration date which was 6 months after preparation day (Frozen).
  Fecal Microbiota: Fecal Microbiota will be delivered via colonoscopy.
- Fecal Microbiota_Lyophilized: Donor stool (greater than 150 grams) was collected <4 hours prior to the procedure and then mixed in a homogenizer with 1500 milliliters (mL) (1:10 dilution) sterilized 0.9% NaCl in a large sterilized suction canister until a smooth consistency was reached. The suspension was filtered using a coffee filter twice. The microbiota suspension (250 milliliters (mL)) was starting lyophilization process within 30 minutes after completion of stool filtration (Lyophilized). Lyophilized microbiota products were kept at 4 degrees celsius (C) and were used within 6 months after preparation day.
  Fecal Microbiota: Fecal Microbiota will be delivered via colonoscopy.
Period: Overall Study
Arm/Group | Fecal Microbiota_Fresh | Fecal Microbiota_Frozen | Fecal Microbiota_Lyophilized
Started | 27 | 27 | 24
Completed | 25 | 25 | 20
Not Completed | 2 | 2 | 4

BASELINE CHARACTERISTICS:
Population: One patient withdraw from the study before starting the procedure
Groups:
- Fecal Microbiota_Frozen: Donor stool (greater than 150 grams) was collected <4 hours prior to the procedure and then mixed in a homogenizer with 1500 milliliters (mL) (1:10 dilution) sterilized 0.9% NaCl in a large sterilized suction canister until a smooth consistency was reached. The suspension was filtered using a coffee filter twice. The microbiota suspension (250mL) was kept at -80 degrees celsius (C) freezer labeled with ID and expiration date which was 6 months after preparation day (Frozen).
  Fecal Microbiota: Fecal Microbiota will be delivered via colonoscopy.
- Total: Total of all reporting groups
Arm/Group | Fecal Microbiota_Fresh | Fecal Microbiota_Frozen | Fecal Microbiota_Lyophilized | Total
Number analyzed (Participants) | 27 | 27 | 24 | 78
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (20.04) | 63 (13.79) | 59 (19.27) | 63 (17.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 18 | 13 | 52
  Male | 6 | 9 | 11 | 26
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 27 | 27 | 24 | 78
Number of Patients with Inflammatory bowel disease [Count of Participants; unit: Participants] | 7 | 4 | 5 | 16
Number of Patients with Ulcerative Colitis [Count of Participants; unit: Participants] | 6 | 3 | 3 | 12
Number of Patients with Crohn's Disease [Count of Participants; unit: Participants] | 1 | 3 | 3 | 7
Number of Patients used Anti-C. difficile infection (CDI) treatment 6 months before the procedure [Count of Participants; unit: Participants] | 25 | 24 | 24 | 73
duration since last Clostridium difficile infection (CDI) bout in 0.5 month increments [Mean (Standard Deviation); unit: half months] | 2 (2.06) | 2 (1.97) | 2 (1.36) | 2 (1.80)
total number Clostridium difficile infection (CDI) bouts before fecal microbiota transplantation [Mean (Standard Deviation); unit: counts] | 4 (0.87) | 4 (0.93) | 4 (2.24) | 4 (1.35)

OUTCOME MEASURES:

1. Primary Outcome: Safety of Fresh, Frozen or Lyophilized Intestinal Bacteria From Healthy Donors Given by Colonoscopy for Therapy in Subjects With Recurrent C. Difficile Associated Diarrhea (RCDAD) as Assessed by Number of Participants Who Any Adverse Event
Description: Any untoward medical occurrence associated with the use of PRIM-DJ2727 whether or not considered drug related is considered as an adverse event (AE)
Time Frame: 6 months
Population: One subject in the Fecal Microbiota_Fresh group was lost to follow up.
Measure: Count of Participants; unit: Participants
Groups:
- Fecal Microbiota_Fresh: Donor stool (greater than 150 grams) was collected <4 hours prior to the procedure and then mixed in a homogenizer with 1500 mL (1:10 dilution) sterilized 0.9% NaCl in a large sterilized suction canister until a smooth consistency was reached. The suspension was filtered using a coffee filter twice. The microbiota suspension (250mL) was used within 2 hours of preparation (Fresh).
  Fecal Microbiota: Fecal Microbiota will be delivered via colonoscopy.
- Fecal Microbiota_Frozen: Donor stool (greater than 150 grams) was collected <4 hours prior to the procedure and then mixed in a homogenizer with 1500 mL (1:10 dilution) sterilized 0.9% NaCl in a large sterilized suction canister until a smooth consistency was reached. The suspension was filtered using a coffee filter twice. The microbiota suspension (250mL) was kept at -80 C freezer labeled with ID and expiration date which was 6 months after preparation day (Frozen).
  Fecal Microbiota: Fecal Microbiota will be delivered via colonoscopy.
- Fecal Microbiota_Lyophilized: Donor stool (greater than 150 grams) was collected <4 hours prior to the procedure and then mixed in a homogenizer with 1500 mL (1:10 dilution) sterilized 0.9% NaCl in a large sterilized suction canister until a smooth consistency was reached. The suspension was filtered using a coffee filter twice. The microbiota suspension (250mL) was starting lyophilization process within 30 minutes after completion of stool filtration (Lyophilized). Lyophilized microbiota products were kept at 4 C and were used within 6 months after preparation day.
  Fecal Microbiota: Fecal Microbiota will be delivered via colonoscopy.
Arm/Group | Fecal Microbiota_Fresh | Fecal Microbiota_Frozen | Fecal Microbiota_Lyophilized
Number analyzed (Participants) | 26 | 27 | 24
Participants | 15 | 23 | 17
Statistical Analysis 1: Comparison: Fecal Microbiota_Fresh vs Fecal Microbiota_Frozen vs Fecal Microbiota_Lyophilized; Test type: Other; p = 0.157, Chi-squared, Corrected

2. Secondary Outcome: Number of Participants Who Had a Subsequent Bout of C-diff Associated Diarrhea
Description: a subsequent bout of C-diff associated diarrhea was defined as diarrhea, C. difficile toxins positive and using anti-C. difficile antibiotic treatment
Time Frame: 30 days
Population: One subject in the Fecal Microbiota_Fresh group was lost to follow up.
Measure: Count of Participants; unit: Participants
Arm/Group | Fecal Microbiota_Fresh | Fecal Microbiota_Frozen | Fecal Microbiota_Lyophilized
Number analyzed (Participants) | 26 | 27 | 24
Participants | 1 | 3 | 7
Statistical Analysis 1: Comparison: Fecal Microbiota_Fresh vs Fecal Microbiota_Frozen vs Fecal Microbiota_Lyophilized; Test type: Other; p = 0.041, Chi-squared, Corrected

ADVERSE EVENTS:
Time Frame: 6 months
Description: Although 27 started in the Fecal Microbiota_Fresh group, only 26 were indicated as "at risk" because one person in the Fecal Microbiota_Fresh group was lost to follow up.
Groups:
- Fecal Microbiota_Fresh: Donor stool (greater than 150 grams) was collected <4 hours prior to the procedure and then mixed in a homogenizer with 1500 mL (1:10 dilution) sterilized 0.9% NaCl in a large sterilized suction canister until a smooth consistency was reached. The suspension was filtered using a coffee filter twice. The microbiota suspension (250 mL) was used within 2 hours of preparation (Fresh).
  Fecal Microbiota: Fecal Microbiota will be delivered via colonoscopy.
- Fecal Microbiota_Frozen: Donor stool (greater than 150 grams) was collected <4 hours prior to the procedure and then mixed in a homogenizer with 1500 mL (1:10 dilution) sterilized 0.9% NaCl in a large sterilized suction canister until a smooth consistency was reached. The suspension was filtered using a coffee filter twice. The microbiota suspension (250 mL) was kept at -80 C freezer labeled with ID and expiration date which was 6 months after preparation day (Frozen).
  Fecal Microbiota: Fecal Microbiota will be delivered via colonoscopy.
- Fecal Microbiota_Lyophilized: Donor stool (greater than 150 grams) was collected <4 hours prior to the procedure and then mixed in a homogenizer with 1500 mL (1:10 dilution) sterilized 0.9% NaCl in a large sterilized suction canister until a smooth consistency was reached. The suspension was filtered using a coffee filter twice. The microbiota suspension (250 mL) was starting lyophilization process within 30 minutes after completion of stool filtration (Lyophilized). Lyophilized microbiota products were kept at 4 C and were used within 6 months after preparation day.
  Fecal Microbiota: Fecal Microbiota will be delivered via colonoscopy.
Arm/Group | Fecal Microbiota_Fresh | Fecal Microbiota_Frozen | Fecal Microbiota_Lyophilized
All-Cause Mortality (participants affected / at risk) | 0/26 | 1/27 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/26 | 1/27 | 1/24
Other Adverse Events (participants affected / at risk) | 2/26 | 2/27 | 6/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fecal Microbiota_Fresh (N=26) | Fecal Microbiota_Frozen (N=27) | Fecal Microbiota_Lyophilized (N=24)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Colitis and enteritis with cholelithiasis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) — Six days after FMT patient developed acute stomach pain and fever with white blood cell (WBC) 40K. Computed tomography (CT) showed colitis and enteritis with cholelithiasis. Stool was negative for C. difficile toxin.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fecal Microbiota_Fresh (N=26) | Fecal Microbiota_Frozen (N=27) | Fecal Microbiota_Lyophilized (N=24)
gastrointestinal complaints (Gastrointestinal disorders) | 1 (1) | 1 (1) | 5 (5) — gastrointestinal complaints including abdominal cramps, lost appetite, nausea, vomiting
Urinary tract infection (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
blood clot (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) — subject had blood clot rectally

LIMITATIONS AND CAVEATS:
Microbiota analyses was not performed on the subjects with Fecal Microbiota Transplantation (FMT) failure who could not provide four stools. Microbiota was not studied at the species level. Limited sample size of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-15): https://cdn.clinicaltrials.gov/large-docs/92/NCT02318992/Prot_SAP_000.pdf